CLINICAL TRIAL: NCT03898557
Title: Behavioral Commitment and Planning Nudges to Increase HIV Self-testing in South Africa, "Plan and Pledge"
Brief Title: Plan and Pledge, HIV Self-testing in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Wits Reproductive Health and HIV Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1195218
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: HIV self-test kits will be distributed at fixed-point distribution sites in the Tshwane district of South Africa and will be grouped into clusters to randomly receive intervention or control. About 44 clusters with an average of 30 participants per cluster, will be selected for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Experimental): Participants randomized to this arm will receive a card with information to report results via WhatsApp, similar to the existing card used in the STAR program. This card will have a dedicated Usual Care WhatsApp number (different from the existing STAR program numbers).
  Potential self-test recipients will be shown the WhatsApp card and instructed on how to anonymously report use of self-test to the WhatsApp number. Recipients will be instructed to message the WhatsApp number for the following reasons:
  1. So study staff know the self-test recipients used the test and it went ok. 2. So study staff can help the self-test recipients understand the results of the test. 3. If the self-test recipients need support from study staff to access care and services.
  Interventions: Behavioral: Provision of HIV self-test
- Plan and Pledge (Experimental): Participants randomized to this arm will revive the Usual Care WhatsApp card and and a brief template to "make a plan" and "make a pledge" for test completion and results reporting, to take the HIV self-test. The card will include a dedicated Plan and Pledge WhatsApp number.
  Potential self-tester recipients will be shown the WhatsApp card, including Plan and Pledge statements, and will be encouraged by STAR field staff to use the card in their own time to make a plan and sign the pledge as part of receiving the test kit and instructions for how to complete the card. Importantly, testers will be able to keep the card for themselves. There is no expectation to share the plan or the pledge signature with the STAR field staff who distribute self-tests. Field staff will clarify for self-tests recipients that the Plan and Pledge process and card do not change the confidentiality of testing in any way.
  Interventions: Behavioral: Provision of HIV self-test with Commitment and planning prompts

INTERVENTIONS:
Behavioral: Provision of HIV self-test with Commitment and planning prompts — The interventions will use behavioral interventions such as commitment and planning prompts to increase the update of HIV self-testing
  Arms: Plan and Pledge
Behavioral: Provision of HIV self-test — This arm will receive a HIV self-test
  Arms: Usual Care

SUMMARY:
The Plan and Pledge pilot will incorporate behavioral economics approaches (nudges) into the pre-existing STAR self-test fixed-site distribution program, implemented by Wits Reproductive Health and HIV Institute (Wits RHI) at the University of Witwatersrand, Johannesburg, South Africa. The objective of this pilot is to examine the use of commitment strategies to increase uptake of HIV self-testing in South Africa.

DETAILED DESCRIPTION:
This study will use a cluster randomized trial design to test the effectiveness of interventions designed to increase usage of self-test and reporting of results by HIV self-tests recipients. Specifically, this study will examine the use of commitment and planning prompts to increase the uptake of HIV self-testing in the Tshwane district in South Africa. The intervention will build on the implementation procedures of STAR program (HIV Self-Testing Africa). The two arms in the study will be: 1) Usual care, "Promote": A card with information to report results via WhatsApp, similar to the existing card used in the STAR program. with a dedicated Usual care WhatsApp number (different from the existing campaign numbers). 2) Plan and Pledge: A card with the information from the Usual Care card plus a brief template to "make a plan" and "make a pledge" for test completion and results reporting, to take the test. The card will include a dedicated Pledge and Plan WhatsApp number.

Self-test distribution team-day pair will serve as the unit of randomization (i.e. two pairs of STAR field staff will be randomized by arm and by day. Clusters of individuals will receive self-tests at a distribution site from a pair of STAR field staff on an individual day). Computer-generated randomization will be used to assign site-day clusters to the 2 study arms. The study will take place at the STAR community fixed-point distribution sites in Tshwane District, South Africa.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older

Exclusion Criteria:

* Intoxication as this effects the result of the HIV self-test

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1479 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers T, Milkman KL, Volpp KG. Commitment devices: using initiatives to change behavior. JAMA. 2014 May;311(20):2065-6. doi: 10.1001/jama.2014.3485. No abstract available. PMID 24777472
- [Background] Cohen J, Rothschild C, Golub G, Omondi GN, Kruk ME, McConnell M. Measuring The Impact Of Cash Transfers And Behavioral 'Nudges' On Maternity Care In Nairobi, Kenya. Health Aff (Millwood). 2017 Nov;36(11):1956-1964. doi: 10.1377/hlthaff.2017.0537. PMID 29137506
- [Background] Milkman KL, Beshears J, Choi JJ, Laibson D, Madrian BC. Using implementation intentions prompts to enhance influenza vaccination rates. Proc Natl Acad Sci U S A. 2011 Jun 28;108(26):10415-20. doi: 10.1073/pnas.1103170108. Epub 2011 Jun 13. PMID 21670283
- [Derived] Buttenheim AM, Schmucker L, Marcus N, Phatsoane M, Msolomba V, Rhagnath N, Majam M, Venter F, Thirumurthy H. Planning and commitment prompts to encourage reporting of HIV self-test results: A cluster randomized pragmatic trial in Tshwane District, South Africa. PLOS Glob Public Health. 2022 Oct 24;2(10):e0001196. doi: 10.1371/journal.pgph.0001196. eCollection 2022. PMID 36962680

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Field staff were not considered enrolled in this study.
Groups:
- Usual Care: Participants randomized to this arm will receive a card with information to report results via WhatsApp, similar to the existing card used in the STAR program. This card will have a dedicated Usual Care WhatsApp number (different from the existing STAR program numbers).
  Potential self-test recipients will be shown the WhatsApp card and instructed on how to anonymously report use of self-test to the WhatsApp number. Recipients (participants) will be instructed to message the WhatsApp number for the following reasons:
  1. To message study staff, so they know that self-test recipients(participants) used the test and it went ok. 2. So study staff can help the self-test recipients (participants) understand the results of the test. 3. If the self-test recipients (participants) need support from study staff to access care and services.
  Provision of HIV self-test: This arm will receive a HIV self-test
- Plan and Pledge: Participants randomized to this arm will revive the Usual Care WhatsApp card and and a brief template to "make a plan" and "make a pledge" for test completion and results reporting, to take the HIV self-test. The card will include a dedicated Plan and Pledge WhatsApp number.
  Potential self-tester recipients (participants) will be shown the WhatsApp card, including Plan and Pledge statements, and will be encouraged by STAR field staff to use the card in their own time to make a plan and sign the pledge as part of receiving the test kit and instructions for how to complete the card. Importantly, testers will be able to keep the card for themselves. There is no expectation to share the plan or the pledge signature with the STAR field staff who distribute self-tests. Field staff will clarify for self-tests recipients (participants) that the Plan and Pledge process and card do not change the confidentiality of testing in any way.
  Provision of HIV self-test with Commitment and planning prompts: The interventions will use behavioral interventions such as commitment and planning prompts to increase the update of HIV self-testing
Period: Overall Study
Arm/Group | Usual Care | Plan and Pledge
Started | 747 | 731
Completed | 747 | 731
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Participants randomized to this arm will receive a card with information to report results via WhatsApp, similar to the existing card used in the STAR program. This card will have a dedicated Usual Care WhatsApp number (different from the existing STAR program numbers).
  Potential self-test recipients will be shown the WhatsApp card and instructed on how to anonymously report use of self-test to the WhatsApp number. Recipients will be instructed to message the WhatsApp number for the following reasons:
  1. So study staff know the self-test recipients used the test and it went ok. 2. So study staff can help the self-test recipients understand the results of the test. 3. If the self-test recipients need support from study staff to access care and services.
  Provision of HIV self-test: This arm will receive a HIV self-test
- Plan and Pledge: Participants randomized to this arm will revive the Usual Care WhatsApp card and and a brief template to "make a plan" and "make a pledge" for test completion and results reporting, to take the HIV self-test. The card will include a dedicated Plan and Pledge WhatsApp number.
  Potential self-tester recipients will be shown the WhatsApp card, including Plan and Pledge statements, and will be encouraged by STAR field staff to use the card in their own time to make a plan and sign the pledge as part of receiving the test kit and instructions for how to complete the card. Importantly, testers will be able to keep the card for themselves. There is no expectation to share the plan or the pledge signature with the STAR field staff who distribute self-tests. Field staff will clarify for self-tests recipients that the Plan and Pledge process and card do not change the confidentiality of testing in any way.
  Provision of HIV self-test with Commitment and planning prompts: The interventions will use behavioral interventions such as commitment and planning prompts to increase the update of HIV self-testing
- Total: Total of all reporting groups
Arm/Group | Usual Care | Plan and Pledge | Total
Number analyzed (Participants) | 747 | 731 | 1478
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-24 | 395 | 390 | 785
  Age: 25-39 | 305 | 280 | 585
  Age: >= 40 | 46 | 57 | 103
  Age: Not reported | 1 | 4 | 5
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/ Gender: Female | 398 | 365 | 763
  Sex/ Gender: Male | 348 | 361 | 709
  Sex/ Gender: Transgender/Not Reported | 1 | 5 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Africa | 747 | 731 | 1478
Most Recent HIV Test [Count of Participants; unit: Participants]
  Never Tested | 82 | 49 | 131
  0-3 Months | 88 | 81 | 169
  3-12 Months | 372 | 368 | 740
  More than 12 months | 197 | 225 | 422
  Not Reported | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Report of HIV Self-test Result
Description: The percent of self-test recipients who report self-test result on the dedicated WhatsApp number and are HIV positive, by study arm and compared to the standard of care arm of the STAR program
Time Frame: approximately 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Plan and Pledge
Number analyzed (Participants) | 747 | 731
Participants
  Reported | 59 | 63
  Not Reported | 688 | 668

2. Secondary Outcome: Report of Positive HIV Self-test Result
Description: The count of negative:positive test results reported by study arm and compared to the standard of care arm of the STAR program.
Time Frame: approximately 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Plan and Pledge
Number analyzed (Participants) | 59 | 63
Participants
  Negative | 59 | 63
  Positive | 0 | 0

3. Other Pre Specified Outcome: Consent for Follow-up
Description: The percent of self-test recipients who consent to phone/SMS follow-up by study arm and compared to the standard of care arm of the STAR program.
Time Frame: approximately 3 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Complete Follow-up
Description: The percent of self-test recipients who are successfully reached for follow-up by phone about 7 days after receiving the HIV self-test, by study arm and compared to the standard of care arm of the STAR program
Time Frame: approximately 3 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: On-site Testing
Description: Percent of on-site testers by study arm and compared to the standard of care arm of the STAR program.
Time Frame: approximately 3 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Confirmatory Testing
Description: The percent of self-test recipients who seek confirmatory testing by study arm and compared to the standard of care arm of the STAR program.
Time Frame: approximately 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 24 day time period.
Arm/Group | Usual Care | Plan and Pledge
All-Cause Mortality (participants affected / at risk) | 0/747 | 0/731
Serious Adverse Events (participants affected / at risk) | 0/747 | 0/731
Other Adverse Events (participants affected / at risk) | 0/747 | 0/731

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT03898557/Prot_SAP_000.pdf